CLINICAL TRIAL: NCT05718427
Title: Effect of Ayres Sensory Integration Therapy on Sensory, Motor, Cognitive, Behavioral Skills and Social Participation in Children With Attention Deficit Hyperactivity Disorder: Randomized Controlled Trial
Brief Title: Effect of ASI on Sensory, Motor, Cognitive, Behavioral Skills and Social Participation in Children With ADHD
Acronym: ASI-ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Busra Kaplan Kilic, Lecturer, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/44353
Record Dates: First submitted 2022-12-27; First posted 2023-02-08 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Sensory Integration Disorder; Motor Activity; Cognitive Deficit in Attention; Behavior Hyperactive; Emotional Regulation; Social Skills
Keywords: ADHD; Sensory Integration; Motor Performance
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Activity; Spasm; Emotional Regulation; Social Skills

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ayres Sensory Integration Therapy Group (Experimental): Ayres Sensory Integration (ASI) therapy will be applied to children in the intervention group. In the intervention group, Ayres Sensory Integration Therapy will be performed 3 days a week for a total of 10 weeks, 60 minutes each session, in accordance with the Ayres Sensory Integration Fidelity Measure (ASI-FM). A manualized protocol will be followed based on the principles of ASI-FM, Ayres sensory integration.
  Interventions: Behavioral: Ayres Sensory Integration Therapy
- Waiting Group (No Intervention): The children in the control group will be wait just 10 weeks. The second evaluation will be repeated 10 weeks after the first evaluation. In order for the children in the control group to benefit from sensory integration therapy, after a 10-week waiting period, after the result measurements are applied again, Ayres sensory integration therapy will be applied 3 days a week with 60 minutes each session in accordance with the Ayres Sensory Integration Fidelity Measure (ASI-FM).

INTERVENTIONS:
Behavioral: Ayres Sensory Integration Therapy — Ayres sensory integration theory provides evidence from basic and applied science about the ability to receive, sort, process, and make use of the information originating from the body and the environment and perceived by our senses (touch, gravity, body position and movement, sight, smell, hearing, taste). This sensory information goes to the brain, where it is organized and interpreted. As a result, we form a plan of action that allows us to have an adaptive response appropriate for the demands of the environment. A thorough assessment guides the preparation of goals addressing the referring concerns and the recommendations for intervention. Ayres Sensory Integration intervention is provided within the context of professional practice. It is designed to improve sensory perceptual abilities, self-regulation, motor skills, and praxis. In doing so, it supports the client's ability to show improved behavior, learning, and social participation.
  Arms: Ayres Sensory Integration Therapy Group

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is a very common neurodevelopmental disorder in childhood characterized by short attention span, impulsivity and hyperactivity. It is also known that sensory integration problems are seen together with the basic symptoms of ADHD. Studies indicate that children with ADHD have difficulties in perceiving and processing sensory stimuli, and in relation to this, they have difficulty in producing appropriate sensory responses at school, at home and in social environments. However, it was observed that the interventions related to ADHD did not focus on the sensory-motor dimension enough, and focused more on cognitive or social skills. Although current research indicates the presence of sensory integration disorder in children with ADHD, there are no studies showing the effectiveness of sensory integration intervention. Our study was planned to examine the effect of Ayres Sensory Integration intervention on sensory-motor, cognitive, behavioral skills and social participation in children with ADHD. Materials and Methods: After the evaluation, 90 children with ADHD will be included in the study by dividing them into intervention (n=45) and control (n=45) groups by simple randomization method. Ayres Sensory Integration Therapy intervention will be applied to the intervention group for 10 weeks, 3 times a week, with a session duration of 1 hour, while the control group will continue the drug treatment and after a waiting period of 10 weeks, Ayres Sensory Integration Therapy will be applied after the second evaluation. Participants, Sensory Profile (SP), Sensory Integration and Praxis Test (SIPT), Emotion Regulation Checklist (ERC), Stroop Test TBAG Form (Stroop TBAG), Childhood Executive Functions Inventory (CHEXI), Participation and Environment Scale for Children and Adolescents (PEM-CY), Conners Teacher Rating Scale (CTRS), Conners Parent Rating Scale (CPRS), Bruininks-Oseretsky Motor Proficiency Test-2 (BOT-2) and Goal Achievement Scale (GAS) both before and before intervention. and post-group change as well as between-group differences will be evaluated.

DETAILED DESCRIPTION:
Although there are studies in the literature showing the presence of Sensory Integration Disorder (SID) in children with ADHD, most researchers have studied a similar profile, such as sensory modulation disorder, and few have investigated all components of sensory integration (such as sensory perception, praxis). More research is needed to confirm the effects of Ayres Sensory Integration (ASI) therapy in children with ADHD and the possible relationship between SID-based difficulties in activities of daily living and ADHD symptoms. In our study, it was aimed to investigate the effect of Ayres Sensory Integration therapy on sensory, motor, cognitive, behavioral and social participation in children with ADHD in the light of extensive literature and recommendations.

ASI therapy will be applied to the intervention group, and the first assessment will be applied to the control group and the second assessment will be made 10 weeks later. However, after a 10-week waiting period, ASI therapy intervention will be applied after the second evaluation so that the children in the control group can also benefit from the intervention. ASI therapy intervention will be applied for 10 weeks, 3 times a week, with a session duration of 1 hour. Inclusion criteria: Being diagnosed with ADHD according to the DSM-V criteria, taking medication, being between the ages of 6 and 8 and attending school. Exclusion criteria: Having previously received sensory integration therapy, having another diagnosis in addition to the ADHD diagnosis.

In addition to drug therapy, ASI therapy will be applied to children in the intervention group. In the intervention group, ASI therapy will be performed 3 days a week for a total of 10 weeks, 60 minutes each session, in accordance with the Ayres Sensory Integration Fidelity Measure (ASI-FM). A manualized protocol will be followed based on the principles of ASI-FM, Ayres sensory integration.

The children in the control group will be given only drug treatment. The second evaluation will be repeated 10 weeks after the first evaluation. In order for the children in the control group to benefit from sensory integration therapy, after a 10-week waiting period, after the result measurements are applied again, ASI therapy will be applied 3 days a week with 60 minutes each session in accordance with the Ayres Sensory Integration Fidelity Measure (ASI-FM).

ELIGIBILITY:
Inclusion Criteria:

* According to the DSM-V criteria diagnosed with ADHD-C type,
* To be on medication,
* To be between the ages of 6 and 8,
* To attend school.

Exclusion Criteria:

* Having previously received sensory integration therapy,
* Having another diagnosis in addition to the ADHD diagnosis.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-02-18 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Sensory Integration and Praxis Test (SIPT) | SIPT will also be used in the initial and final assessment at week 1 and week 12. SIPT measures the change in sensory skills.Getting a high score on the test means good performance.
  Developed by Ayres, is a standardized performance-based observational test that evaluates sensory perception and sensory perception-based skills in detail in children between the ages of 4 and 8 years and 11 months. SIPT, is one of the important gold tests in evaluating sensory development.
Bruininks-Oseretsky Motor Proficiency Test-2 (BOT-2) | BOT-2 will also be used in the initial and final assessment at week 1 and week 12. BOT-2 measures the change in motor skills. Getting a high score on the test means good performance.
  Bruininks-Oseretsky Motor Proficiency Test-2 (BOT-2) is a test developed for children aged 4-21 and developed to measure the motor functions of children. BOT-2 is an observational assessment evaluating motor performance, consisting of 8 subtests and 12 items in total. It consists of fine motor accuracy, fine motor integration, dexterity, bilateral coordination, balance, upper extremity coordination, endurance, speed and agility subtests.
Goal Attainment Scale (GAS) | GAS will also be used in the initial and final assessment at week 1 and week 12. GAS measures the change in behavior. Maximum +2 and minimum -2 points are taken. +2 means the best result.
  The Goal Attainment Scale (GAS) is used to evaluate the achievement of functional therapy goals in children receiving treatment in pediatric services. It helps to set priorities and clear goals for intervention. It provides the child's continuous interest in the set goals and offers a person-centered approach. The determined goals should be specific, measurable, achievable, relevant and well-timed. While applying GAS, goals are set for the child and possible outcomes are defined for each goal. After a certain intervention, the functional status of the child is determined again. GAS consists of 5 points as -2, -1, 0, +1 and +2. A score of -2 indicates the child's pre-intervention baseline level, a score of -1 indicates a development below the expected attainment level, a score of 0 indicates an expected attainment level, a score of +1 indicates a better-than-expected achievement, and a score of +2 indicates that the child performs much better than expected.

SECONDARY OUTCOMES:
Emotional Regulation Checklist (ERC) | ERC will also be used in the initial and final assessment at week 1 and week 12. The test provides subjective data about emotional regulation behaviour in child. Getting a high score on the test means good performance.
  The Emotional Regulation Checklist (ERC) is a 24-item scale developed by Shields and Cicchetti to evaluate the emotion regulation competence of children aged 6-13 and can be evaluated by both parents and teachers.
Childhood Executive Functions Inventory (CHEXI) | CHEXI will also be used in the initial and final assessment at week 1 and week 12. The test provides subjective data about executive functions skills in child. Getting a high score on the test means good performance.
  Childhood Executive Functions Inventory (CHEXI) is a scale consisting of 26 questions for children aged 4-12 years, developed by Lisa B. Thorell and Lilianne Nyberg as a measurement focusing especially on executive functions.
Participation and Environment Scale for Children and Youth (PEM-CY) | PEM-CY will also be used in the initial and final assessment at week 1 and week 12. The test provides subjective data about participation area in child. Getting a high score on the test means good performance.
  The Participation and Environment Scale for Children and Youth (PEM-CY) is a 28-item questionnaire assessing participation in children aged 5-17 years. It is a family-reported scale that questions the child's participation in school, home and society.
Stroop Test TBAG Form (Stroop TBAG) | Stroop TBAG will also be used in the initial and final assessment at week 1 and week 12. Stroop TBAG measures the change in cognitive skills. Getting a high score on the test means good performance.
  The Stroop Test TBAG Form (Stroop TBAG) is one of the golden tests used to measure selective attention and ability to shift attention, focusing on the color used in the spelling of the word and the disruptive effect of the color in the pronunciation of the word.

OTHER OUTCOMES:
Sensory Profile (SP) | SP will also be used in the initial and final assessment at week 1 and week 12. The test provides subjective data. The results are interpreted as exact difference, probable difference and typical performance.
  The Sensory Profile (SP) is a family-reported scale that provides data on children's reactions to sensory events in daily life, how sensory behaviors can contribute to performance in daily life, and what difficulties they cause in performance. It consists of 125 questions that can be applied between the ages of 3-10.
Conners Parent Rating Scale (CPRS) | CPRS will also be used in the initial and final assessment at week 1 and week 12. The test provides subjective by parent data about child general behaviour. Getting a high score on the test means good performance.
  Conners Parent Rating Scale (CPRS) is important behavioral screening and diagnostic scales that have a wide range between the ages of 3-17 and are used quite frequently especially in ADHD. CPRS consists of 48 items developed to child behavior.
Conners Teacher Rating Scale (CTRS) | CTRS will also be used in the initial and final assessment at week 1 and week 12. The test provides subjective by teacher data about child school behaviour. Getting a high score on the test means good performance.
  Conners Teacher Rating Scale (CTRS) is important behavioral screening and diagnostic scales that have a wide range between the ages of 3-17 and are used quite frequently especially in ADHD. CTRS consists of 28 items developed to grade students' classroom behaviors by their teachers.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT05718427/Prot_SAP_000.pdf